CLINICAL TRIAL: NCT02529267
Title: Prospective Abuse and Intimate Partner Violence Surgical Evaluation (PRAISE-2) : A Multicentre Pilot Prospective Cohort Study
Brief Title: Prospective Abuse and Intimate Partner Violence Surgical Evaluation
Acronym: PRAISE-2
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: PRAISE-2
Record Dates: First submitted 2015-08-07; First posted 2015-08-20 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Fractures, Bone; Dislocations; Spouse Abuse
Keywords: Cohort Studies; intimate partner violence; orthopaedic surgery; epidemiology; outcomes in fracture care
MeSH Terms: conditions — Fractures, Bone; Joint Dislocations | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Experienced abuse: Experienced IPV in the past 12 months
  Interventions: Other: Standard of care
- Did not experience abuse: Did not experience IPV in the past 12 months.
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: Standard of care

SUMMARY:
Intimate partner violence (IPV), also known as domestic abuse, is a leading cause of non-fatal injury in women worldwide. 1 in 6 women attending surgical fracture clinics have a history of IPV in the past year. Given the high prevalence and costs associated with IPV, there is a need to identify health outcomes associated with IPV, the incidence of new and worsening cases of IPV, and resource use among IPV victims. This prospective cohort study of women with fractures and dislocations will assess differences in injury-related outcomes (time to fracture healing, injury-related complications, and return to pre-injury function) between abused and non-abused women. This study will also determine whether a musculoskeletal injury can lead to new or worsening abuse by an intimate partner and how patterns of IPV change over time following musculoskeletal injuries.Finally, the proposed study will also inform the feasibility of a larger multinational cohort study.

DETAILED DESCRIPTION:
Number of Participants:

250

Primary Research Objectives:

Feasibility

Secondary Research Objective:

The secondary objectives are to determine:

1. How a history of IPV affects injury-related complications;
2. How a history of IPV affects return to pre-injury function;
3. Incident cases of IPV after a musculoskeletal injury, if the injury was not the result of IPV;
4. How a history of IPV affects health care and support service use after a musculoskeletal injury;
5. How a history of IPV affects health-related quality of life after a musculoskeletal injury;
6. How patterns of IPV change over time after a musculoskeletal injury;
7. How abused women's stage of change changes over time after a musculoskeletal injury

Diagnosis and Main Inclusion Criteria:

The inclusion criteria are:

1. adult females (at least 16 or 18 years of age depending on local ethics requirements);
2. patients presenting to participating fracture clinics within 6 weeks of their musculoskeletal injury;
3. patients presenting with a fracture or dislocation which is being managed with either surgical or non-surgical treatment.

The exclusion criteria are:

1. unwilling to or unable to provide consent;
2. unable to complete the study questionnaires in a private location, due to safety and confidentiality;
3. unwilling or unable to follow the study protocol or their attending surgeon has concerns about their ability or willingness to follow study protocols;
4. does not speak and write in English or the dominant language of the local clinic

Study Outcomes:

The primary outcome is feasibility. Secondary outcomes are injury-related complications, return to function, incidence of IPV, quality of life, abuse type and severity, and stage of change.

Duration of Patient Follow-Up:

Study participants will be followed for 12 months

ELIGIBILITY:
Inclusion Criteria:

* Adult females
* Patients presenting to participating fracture clinics within 6 weeks of their musculoskeletal injury
* Patients presenting with a fracture or dislocation which is being managed with either surgical or non-surgical treatment

Exclusion Criteria:

* Unwilling to or unable to provide consent
* Unable to complete the study questionnaires in a private location
* Unwilling or unable to follow the study protocol or their attending surgeon has concerns about their ability or willingness to follow study protocols
* Does not speak and write in English or the dominant language of the local clinic

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult women presenting to participating fracture clinics with a fracture or dislocation.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2015-08; Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility - Recruitment rate | 12 months
  Number of patients recruited at each site during a 12 month period
Feasibility - Proportion of Missed and/or out of window visits | 12 months
  Proportion of missed and out of window visits
Feasibility - Collection of secondary outcomes (Proportion of included patients followed at 12 months for the primary and secondary outcomes) | 12 months
  Proportion of included patients followed at 12 months for the primary and secondary outcomes
Feasibility - Completion of data collection (proportion of case report forms, including patient questionnaires, completed at 12 months) | 12 months
  The proportion of case report forms, including patient questionnaires, completed at 12 months.

SECONDARY OUTCOMES:
Proportion of patients with injury-related complications assessed by central adjudication | 12 months
  Compare proportion of patients experiencing a composite of injury-related complications between patients who self-report a history of IPV and those who do not. Injury-related complications include non-union, malunion, infection, unplanned secondary procedure, mortality, hardware failure, etc. An independent, blinded adjudicator will determine whether the event is injury-related.
Return to function questionnaire | 12 months
  We will use the Return to Function Questionnaire (RTF) to compare the mean time to return to pre-injury function among women who disclose a history of IPV versus those who do not disclose IPV. The RTF is a 4 question tool that was used in a recently completed large FDA-regulated fracture trial.
IPV incidence questionnaire | 12 months
  Women's self-reported experience of IPV will be measured using a direct method of screening used by the PRAISE Investigators in 2 previous studies conducted in trauma populations. A participant will be considered to have disclosed IPV if she answers positively to at least 1 of the 3 direct screening questions.
Resource use questionnaire | 12 months
  Women's access to and use of health and support services will be measured by directly asking participants to self-report if they have accessed health care services, a social worker, mental health professional, women's shelter, helpline, violence against women website, or legal assistance.
Quality of life - EQ-5D | 12 months
  Participants' quality of life will be measured using the EuroQol-5 Dimensions (EQ-5D), a widely used and well-validated quality of life tool. The EQ-5D is a comprehensive, 5-item compact health status classification and health state preference questionnaire.
IPV frequency questionnaire | 12 months
  Using 3 questions from the Woman Abuse Screening Tool, which categorizes frequency of different types of violence, we will record and analyze changes in frequency of IPV experienced over time.
Stage of change questionnaire | 12 months
  Participants will complete the Domestic Violence Survivor Assessment (DVSA) Short Form questionnaire to determine her stage of change. The stages of change are based on the transtheoretical model of health behavior change applied specifically to survivors of abuse. We developed the DVSA Short Form for the purpose of this study, with the aim of making the self-administered form more accessible.
IPV type questionnaire | 12 months
  Using 3 questions from the Woman Abuse Screening Tool, which categorizes types of violence as physical, emotional, and/or sexual abuse, we will record and analyze changes in type of IPV experienced over time.

CONTACTS AND LOCATIONS:
Overall Officials: Brad Petrisor, MD, MSc, Principal Investigator — Hamilton Health Sciences Corporation; Sheila Sprague, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

REFERENCES:
- [Background] PRAISE Investigators; Sprague S, Bhandari M, Della Rocca GJ, Goslings JC, Poolman RW, Madden K, Simunovic N, Dosanjh S, Schemitsch EH. Prevalence of abuse and intimate partner violence surgical evaluation (PRAISE) in orthopaedic fracture clinics: a multinational prevalence study. Lancet. 2013 Sep 7;382(9895):866-76. doi: 10.1016/S0140-6736(13)61205-2. Epub 2013 Jun 12. PMID 23768757
- [Derived] Madden K; PRAISE-2 Investigators. Prospective evaluation of intimate partner violence in fracture clinics (PRAISE-2): protocol for a multicentre pilot prospective cohort study. Pilot Feasibility Stud. 2018 Jun 15;4:115. doi: 10.1186/s40814-018-0301-9. eCollection 2018. PMID 29946480